CLINICAL TRIAL: NCT04642612
Title: Cerebral Blood Flow Evaluation With Trancranial Doppler After Unilateral Interscalene Nerve Block: Observational Prospective Study
Brief Title: Cerebral Blood Flow Evaluation With Trancranial Doppler After Interscalene Nerve Block
Acronym: CBF-TCD
Status: Terminated | Type: Observational
Why Stopped: Study not properly designed for outcome measure
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Anna Maria Bombardieri, Clinical Assistant Professor of Anesthesiology, Perioperative and Pain Medicine, Stanford University, Stanford University
Other Study IDs: 59007
Record Dates: First submitted 2020-11-02; First posted 2020-11-24 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Regional Anesthesia; Horner Syndrome; Cerebral Blood Flow
MeSH Terms: conditions — Horner Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Treatment Arm: Patients ages 18-85 years old presenting with orthopedic shoulder surgery with indication to receive preoperative insertion of interscalene nerve block.
  Interventions: Device: TCD Measurement

INTERVENTIONS:
Device: TCD Measurement — CBFV measurements will be acquired continuously with the patient supine and the head neutral. Analysis of CBFV measurements will be undertaken at 3 timepoints:
  1. Patient awake and supine in the holding area
  2. After sedation
  3. After interscalene nerve block

SUMMARY:
The purpose of this study is to assess cerebral blood flow velocity (CBFV) following regional anesthesia for shoulder surgery. The results of this study will help to further understand the physiologic effect of the interscalene nerve block on cerebral blood flow.

DETAILED DESCRIPTION:
Traditionally, cerebral blood flow (CBF) is believed to decline when mean arterial pressure (MAP) is below the lower limit of cerebral autoregulation. Cerebral blood flow autoregulation refers to the capacity of the central nervous system to maintain blood flow within a wide range of mean arterial blood pressure.

The habitual thinking is that the brain is perfused merely dependent by the blood pressure and that above or below the limits of cerebral autoregularion CBF is pressure passive. Despite this notion, there is evidence showing that parameters other than MAP influence cerebral hemodynamics independent of cerebral autoregulation. One of the physiologic processes that contribute to CBF regulation is cardiac output (CO). However, exactly how an alteration in CO, in the face of a stable blood pressure, leads to a change in CBF is not entirely clear.

One of the suggested mechanisms in play is the sympathetic nervous system (SNS)-mediated vasoconstriction of extracranial and proximal intracranial vessels. Cerebral arteries are abundantly innervated by sympathetic nerve fibers originating from the superior cervical ganglion. Studies have shown that CBF reduction is attenuated by pharmacologic blockade or extirpation of the cervical sympathetic chain.

The anesthetic protocol for patients undergoing major shoulder surgery include an interscalene nerve block (ISNB) combined with general anesthesia in the sitting position. The ISNB involves injecting local anesthetic at the level of the cervical spinal roots. One of the most common side effects encountered after ISNB is Horner syndrome, which is characterized by ptosis, myosis, and enopthalmia. Horner's syndrome results from the diffusion of the local anesthetic solution to the ipsilateral sympathetic cervical chain (stellate ganglion). The presence of Horner's syndrome indicates spread of local anesthetic to the sympathetic chain.

Whether this degree of sympatholytic following interscalene block is associated with an observable change in CBF is unknown. Studies in baboon have shown that cervical surgical sympathectomy maintained CBF in the face of hemorrhagic hypotension and CBF did not decrease until MAP was 35% of the baseline value. These results suggest that sympathectomy induced by the block of the sympathetic chain by the local anesthetic injected for the ISNB might alter CBF. Therefore, the aim of our study is to evaluate the effect of unilateral interscalene nerve block on CBF by measuring CBF velocity non-invasively with Transcranial doppler (TCD).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing orthopedic surgery and with an indication for preoperative insertion of interscalene nerve block
* 18-85 years old
* Give consent to participate in study

Exclusion Criteria:

* Cannot give consent
* Patients who are clinically unstable or require urgent/emergent intervention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing orthopedic surgery with an indication for preoperative insertion of interscalene nerve block, aged 18-85 years old, and give consent to participating in study.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
Cerebral Blood Flow Velocity before and after interscalene nerve block | baseline, after 30 minutes
  The TCD automatically measures blood flow velocity in the main cerebral arteries of the circle of Willis. We will target the MCA which is the closest to the temporal bone therefore the most easily accessible for insonation and monitoring. We will do a bilateral monitoring.

SECONDARY OUTCOMES:
Systolic, diastolic, mean blood pressure changes before and after interscalene nerve block | baseline, after 30 minutes
  Will be measured before/during/after interscalene nerve block placement
Heart Rate | baseline, after 30 minutes
  Will be measured before/during/after interscalene nerve block placement
Respiratory Rate changes before and after interscalene nerve block | baseline, after 30 minutes
  Will be measured before/during/after interscalene nerve block placement
EtCO2 changes before and after interscalene nerve block | baseline, after 30 minutes
  Will be measured before/during/after interscalene nerve block placement
SpO2 changes before and after interscalene nerve block | baseline, after 30 minutes
  Will be measured before/during/after interscalene nerve block placement
Type of local anesthetic | 30 minutes after the nerve block
  Local anesthetic characteristics will be collected after interscalene block placement.
Position of the needle on the cervical trunk for interscalene nerve block | Baseline
  Needle position for interscalene nerve block insertion will be assessed at the time of interscalene block placement
Volume of of local anesthetic | 30 minutes after the nerve block
  Local anesthetic characteristics will be collected after interscalene block placement.
Concentration of local anesthetic | 30 minutes after the nerve block
  Local anesthetic characteristics will be collected after interscalene block placement.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Maria Bombardieri, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Background] Meng L, Hou W, Chui J, Han R, Gelb AW. Cardiac Output and Cerebral Blood Flow: The Integrated Regulation of Brain Perfusion in Adult Humans. Anesthesiology. 2015 Nov;123(5):1198-208. doi: 10.1097/ALN.0000000000000872. PMID 26402848
- [Background] Drummond JC. Cardiac Output: The Neglected Stepchild of the Cerebral Blood Flow Physiology Family. J Neurosurg Anesthesiol. 2020 Apr;32(2):93-94. doi: 10.1097/ANA.0000000000000677. No abstract available. PMID 31972625
- [Background] ter Laan M, van Dijk JM, Elting JW, Staal MJ, Absalom AR. Sympathetic regulation of cerebral blood flow in humans: a review. Br J Anaesth. 2013 Sep;111(3):361-7. doi: 10.1093/bja/aet122. Epub 2013 Apr 24. PMID 23616589
- [Background] Fitch W, MacKenzie ET, Harper AM. Effects of decreasing arterial blood pressure on cerebral blood flow in the baboon. Influence of the sympathetic nervous system. Circ Res. 1975 Nov;37(5):550-7. doi: 10.1161/01.res.37.5.550. PMID 153
- [Background] Seltzer JL. Hoarseness and Horner's syndrome after interscalene brachial plexus block. Anesth Analg. 1977 Jul-Aug;56(4):585-6. doi: 10.1213/00000539-197707000-00033. No abstract available. PMID 560150